CLINICAL TRIAL: NCT02983149
Title: A Clinical Comparison of Two New Bronchial Blockers vs. Double Lumen Tubes in One Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Manager Anesthesia Research, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-7478-A
Record Dates: First submitted 2016-04-14; First posted 2016-12-06 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Thoracic Surgery, Lung Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Double lumen tube (Other): One lung ventilation will be achieved using a double lumen tube
  Interventions: Device: Double lumen tube
- Fuji blocker (Other): One lung ventilation will be achieved using the Fuji blocker
  Interventions: Device: Fuji blocker
- EZ blocker (Other): One lung ventilation will be achieved using the EZ blocker
  Interventions: Device: EZ blocker

INTERVENTIONS:
Device: Double lumen tube — Use an double lumen tube to achieve one lung ventilation in thoracic surgeries
  Arms: Double lumen tube
Device: Fuji blocker — Use the Fuji blocker to achieve one lung ventilation in thoracic surgeries
  Arms: Fuji blocker
Device: EZ blocker — Use the EZ blocker to achieve one lung ventilation in thoracic surgeries
  Arms: EZ blocker

SUMMARY:
Patients undergoing thoracic surgery require selective ventilation of one lung, which allows surgery to proceed on the operative lung that is deflated, and no longer moving. One-lung ventilation (OLV) may be achieved by the use of a double lumen endotracheal tube (DLT) or the placement of a bronchial blocker (BB) via a single lumen endotracheal tube, both of which are in routine clinical use at University Health Network.

Recently, the Endobronchial Blocker (EZ blocker) has been marketed, with a forked tip design and two balloons, one of which is designed to fall into each of the right and left sides, it may require less repositioning. Initial clinical experience with the EZ Blocker suggests that it may be less likely than other blockers to become malpositioned during surgery.

This study will compare the EZ blocker to the Fuji blocker, the most frequently used blocker at this institution, and to double-lumen tubes, the most commonly used devices to provide lung isolation, with respect to intra-operative malpositioning and the speed of lung separation and efficacy of lung collapse during thoracic surgery.

Patients will be randomly assigned, to one of the three study groups: EZ Blocker, Fuji, or left-sided DLT, immediately prior to induction of anesthesia.

The primary end points of time to lung isolation and number of required repositioning maneuvers.

DETAILED DESCRIPTION:
STUDY END POINTS The time required to achieve lung separation, from beginning of laryngoscopy to lung isolation (inflation of the bronchial cuff or blocker), will be recorded. The thoracic surgeons, using a verbal analogue scale, will assess the lung collapse(lung collapse scores-LCS, 0=no collapse, to 10=complete collapse). The LCS will be assessed and recorded as they open the pleura during the procedure (LCS 0), and at 10 min., (LCS 10), and 20 min. (LCS 20) after opening the pleura. The surgeons will be blinded to the lung isolation device used in the patient. If the lung collapse is not satisfactory, the FOB will be passed to assess the lung isolation, and if necessary reposition the device. A malposition will be defined as a clinically obvious relocation of the devise in the trachea or bronchus and a loss of lung isolation interfering with surgery. The number of repositions of the lung isolation device after initial supine placement, airway pressures, tidal volumes, duration of surgery, and the arterial blood gases 20 minutes after pleural opening will be noted.

In addition to the primary end points of time to lung isolation and number of required repositioning maneuvers, the following variables will be recorded: Age, gender, weight, height, BMI, ASA, airway Mallampati score, pulmonary spirometry (if clinically performed: TLC, FEV1, FVC, DLCO), LCS 0/10/20, ventilatory parameters on OLV (airway pressure, tidal volume, respiratory rate, compliance, duration of OLV and surgery, arterial blood gas 20 minutes after opening the pleura (pH, paO2, pCO2 bicarbonate, base excess, oxygen saturation), and finally the dimensions of the left main bronchus (LMB) and the right main bronchus (RMB) using the on-screen program of the radiology server on the pre-operative chest imaging, by the anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Thoracic surgery requiring one-lung ventilation for > 30 minutes.
* Able to provide first party consent.

Exclusion Criteria:

* Known prior difficult intubation.
* Upper airway exam suggestive of difficult intubation.
* Surgical procedure requiring a right double lumen endotracheal tube (such as left pneumonectomy).
* Evidence on clinically required radiologic imaging of abnormal lower airway anatomy, such as right upper lobe origin of the bronchus.
* Prior thoracic surgery or pleurodesis of the operative side (would delay lung collapse).
* History of severe restrictive lung disease (such as pulmonary fibrosis or emphysema) which may affect inflation/deflation times.
* Trauma patients requiring video-assisted thoracoscopic surgery
* Has condition(s) that contraindicate a double lumen endotracheal tube (DLT) or the placement of a bronchial blocker (BB) via a single lumen endotracheal tube.
* Patients with communication difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Time required for lung separation | From initial laryngoscopy to lung isolation will be measured for 0 hours (procedure start) to 3 hours (procedure end time)
  The time required to achieve lung separation, from beginning of laryngoscopy to lung isolation.
Number of repositioning maneuvers of the device | After initial patient's supine position for the duration of the operation 0-3 hours will be recorded
  The number of repositions of the lung isolation device after initial supine placement
Lung collapse scores | The thoracic surgeons, using a verbal analogue scale, will be assessing the lung collapse score (LCS), from 0=no collapse to 10=complete collapse. LCS will be assessed just after opening the pleura, at 10 min., and 20 min. after opening the pleura.
  Time Frame: After opening the pleura, the lung collapse scores will be measured at 0, 10 and 20 minutes (from pleura opening)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Slinger, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, 200 Elizabeth St., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No